CLINICAL TRIAL: NCT05337813
Title: Effects of Low-intensity Excoporeal Shock Wave Therapy (LiESWT) on Women With Pelvic Floor Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KMUHIRB-F(I)-20200050
Record Dates: First submitted 2022-03-21; First posted 2022-04-20 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Overactive Bladder; Stress Incontinence; Interstitial Cystitis; Female Sexual Dysfunction
Keywords: LiESWT
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Stress; Cystitis, Interstitial

STUDY DESIGN:
Intervention Model Description: Only one arm for each disease (LiESWT group)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A. Overactive bladder (Experimental): Overactive bladder (LiESWT therapy once a week, duration 8 weeks)
  Interventions: Device: "Storz Medical" Extracoporeeal Shock Wave Therapy System
- B. Stress incontinence (Experimental): Stress incontinence (LiESWT therapy once a week, duration 8 weeks + PRP therapy once a month, duration 3 months)
  Interventions: Device: "Storz Medical" Extracoporeeal Shock Wave Therapy System
- C. Interstitial cystitis (Experimental): Interstitial cystitis (LiESWT therapy once a week, duration 8 weeks + PRP therapy once a month, duration 3 months)
  Interventions: Device: "Storz Medical" Extracoporeeal Shock Wave Therapy System
- D. Female sexual dysfunction (Experimental): Female sexual dysfunction (LiESWT therapy once a week, duration 8 weeks)
  Interventions: Device: "Storz Medical" Extracoporeeal Shock Wave Therapy System

INTERVENTIONS:
Device: "Storz Medical" Extracoporeeal Shock Wave Therapy System — A. B. C. D. groups need to Low Energy Extracorporeal Shock Wave (LiESWT) therapy once a week, duration 8 weeks(B.、C. groups needs to be combined PRP treatment at 1, 5, 9 weeks)
  Other Names: AEON PRP: APA-15

SUMMARY:
1. This study needles female reproductive urinary tract, likely bladder hyperactivity, active urinary incontinence and interstitial cystitis, observation use of low-capacity seismic wave (LiESWT) therapy combined with combined platelet plasma (PRP), improved bone basin pain and female Urinary incontinence.
2. LiESWT to arousal the clitoris angiogenesis to prevent female sexual dysfunction.

DETAILED DESCRIPTION:
Collect 120 women(A. Overactive bladder、B. Stress incontinence、C. Interstitial cystitis D. Female sexual dysfunction), Low Energy Extracorporeal Shock Wave (LiESWT) therapy once a week, duration 8 weeks(B.、C. PRP treatment at 1, 5, 9 weeks), and to complete all treatment after 4 weeks and 24 weeks back to the clinic, evaluation questionnaire (OABSS、UDI-6、IIQ-7、ICIQ-SF、POPDI-6、FSFI)、Urinary tract dynamics test、Urination log、Cotton pad test、Blood test(ESR、CA125、CBC、CRP). ○DLow Energy Extracorporeal Shock Wave (LiESWT) therapy once a week, duration 4 weeks, and to complete all treatment 4th and after 4 weeks back to the clinic, Pelvic Doppler ultrasound ,evaluation questionnaire (OABSS、UDI-6、IIQ-7、ICIQ-SF、POPDI-6、FSFI).

ELIGIBILITY:
Inclusion Criteria:

1. One of the following symptoms can be included:

   1. Overactive bladder
   2. Stress incontinence
   3. Interstitial cystitis
   4. Not Menopause and female sexual dysfunction (FSFI scores< 26)
2. The blood test confirmed that the number of platelets was 150,000 to 450,000 / UL, and the coagulation function (PT) index was normal.
3. Women over 20 years.

Exclusion Criteria:

1. No UTI during the past week.
2. Patients with poorly controlled diabetes, spinal cord injury, brain disease and neurogenic disease.
3. urinary symptoms of inflammation(Bladder stones、hematuria、urethral syndrome).
4. Patients with acute or chronic infectious diseases.
5. Patients with acute or chronic cardiovascular disease.
6. Patients with a history of chronic liver and kidney disease.
7. Patients receiving anticoagulant therapy(Aspirin and NSAIDs COX-1).
8. Patients with bleeding disorders.
9. Receive low energy extracorporeal shock wave treatment within 1 month before entering the trial.
10. Urinary incontinence need to install the catheter.
11. Pregnant women.
12. Unable to sign the consent form.

Ages: 20 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — women with pelvic floor dysfunction
Enrollment: 120 (Estimated)
Dates: Start 2020-04-10 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Reduce bladder leakage and symptoms of overactive bladder, including urgency, incontinence and nocturia. | 8 months
  1.Questionnaire assessment before and after treatment (OABSS, UDI-6, IIQ-7, ICIQ-SF, POPDI-6, FSFI) . 2.urodynamic examination before and after treatment
Assess the patient for changes in lower abdominal pain | 8 months
  VAS pain index record before and after treatment

SECONDARY OUTCOMES:
Promote the repair and proliferation of blood vessels in the vulva to improve sexual function and improve the overall quality of sexual life. | 2 months
  Doppler ultrasound of the vulva to record the degree of blood congestion before and after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital (KMUH), Kaohsiung City, Sanmin Dist, Taiwan

IPD SHARING:
Plan to Share IPD: No